CLINICAL TRIAL: NCT01799707
Title: Vision Restoration Training in Glaucoma - A Double-blind, Randomized, Placebo-controlled Clinical Trial
Brief Title: Vision Restoration Training in Glaucoma
Acronym: gVRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Magdeburg (Other)
Responsible Party: Principal Investigator, Bernhard A. Sabel, Director, Principle Investigator and Study Director, University of Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VRT 03-2003
Record Dates: First submitted 2013-02-21; First posted 2013-02-27 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Glaucoma
Keywords: vision; restoration; visual field
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vision restoration training (Active Comparator): Vision restoration training (VRT): visual stimuli repetitively presented to stimulate areas of residual vision. The training consists of luminance increment stimuli similar to perimetry and the task isa simple detection task (pressing a key whenever a target stimulus was detected).
  Interventions: Behavioral: vision restoration training
- Discrimination training (Placebo Comparator): Discrimination training. Here, the stimulus is a line segment (bar) which is always presented within the central ±5° visual field in one of four possible random orientations: horizontal, vertical, oblique to the right or oblique to the left. If the patient has visual field defects in this central area, 80% of the stimuli are presented in the intact part of the training region. The task is to identify the orientation of the line segment and press, as fast as possible, one of 4 assigned buttons on the keyboard.
  Interventions: Behavioral: Discrimination Training

INTERVENTIONS:
Behavioral: vision restoration training — visual stimuli repetitively presented to stimulate areas of residual vision. The training consists of luminance increment stimuli similar to perimetry and the task isa simple detection task (pressing a key whenever a target stimulus was detected).
  Other Names: gVRT
  Arms: vision restoration training
Behavioral: Discrimination Training — the stimulus is a line segment (bar) which is always presented within the central ±5° visual field in one of four possible random orientations: horizontal, vertical, oblique to the right or oblique to the left. If the patient has visual field defects in this central area, 80% of the stimuli are presented in the intact part of the training region. The task is to identify the orientation of the line segment and press, as fast as possible, one of 4 assigned buttons on the keyboard.
  Arms: Discrimination training

SUMMARY:
Importance: Visual field loss after retinal damage in glaucoma is considered irreversible and methods are needed to achieve vision restoration. Behavioral vision restoration training (VRT), shown to improve visual fields in hemianopia and optic nerve damage, might comprise such a method.

Objective: To determine if behaviorally activating areas of residual visual (ARV) using VRT by daily one hour training for 3 months improves detection performance in perimetry compared to a vision discrimination task in the intact visual field sector.

DETAILED DESCRIPTION:
Design: Prospective, randomized, double-blind, placebo controlled trial. Setting: Ambulatory care and home training Participants: Volunteer sample of glaucoma patients (25-80 yrs old) with stable visual fields and well controlled intraocular pressure (IOP).

Intervention: Computer-based home training with VRT (n=15) or placebo discrimination training (n=15).

Main Outcome Measures: The primary endpoint is change in detection performance in High Resolution Perimetry (HRP). Secondary endpoints are 30° white/white and 30° blue/yellow near-threshold perimetry. Further measures are eye movements, vision-related quality of life (vQoL) as assessed with (NEI-VFQ) and health-related quality of life (hQoL) using SF-36 Health Survey-Short Form.

Investigators hypothesize that VRT will improve visual performance in glaucoma

ELIGIBILITY:
Inclusion Criteria:

* Visual filed defect caused by glaucoma
* Presence of a reproducible and stable visual field defect inside 30° eccentricity in at least one eye in 2 consecutive ophthalmologic visits during the last 12 months before recruitment
* Well controlled intraocular pressure (IOP), and (iv) age between 25 and 80 years

Exclusion Criteria:

* History of any medical condition precluding scheduled study visits or completion of the study (e.g. unstable cardiovascular disease)
* History of any chronic degenerative or chronic inflammatory disease that could affect the visual field (e.g. multiple sclerosis, tumor
* History of trauma or any non-glaucoma ocular diseases (e.g. diabetic retinopathy, age-related macular degeneration, macular detachment, vascular occlusion
* Severe cognitive or motor impairments
* Insufficient fixation ability
* Photosensitivity
* Intraocular surgery or laser treatment performed within the previous 12 months before recruitment; OR
* Scheduled intraocular surgery

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-07; Primary Completion 2007-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Detection accuracy change in percent over baseline of the visual field | between baseline and 3 months of training
  visual stimulus detection in residual and absolutely defect field of vision will be assessed using computer-based high resolution perimetry (HRP)

SECONDARY OUTCOMES:
change in visual stimulus perimetric detection rate | between baseline and 3 months of training
  improvement of visual field in near-threshold perimetry measured by static perimetry (average threshold in db, average excentricity in degrees of visual angle
improvement of reaction time | between baseline and 3 months of training
  change in average reaction time in ms, measured by HRP

OTHER OUTCOMES:
Eye movement control | between baseline and 3 months of training
  visual stimulus detection in residual and absolutely defect field of vision will be assessed using computer-based high resolution perimetry (HRP)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard A Sabel, PhD, Principal Investigator — University of Magdeburg

REFERENCES:
- [Derived] Sabel BA, Gudlin J. Vision restoration training for glaucoma: a randomized clinical trial. JAMA Ophthalmol. 2014 Apr 1;132(4):381-9. doi: 10.1001/jamaophthalmol.2013.7963. PMID 24504128